CLINICAL TRIAL: NCT01977313
Title: Genetic Polymorphism of the Androgen Receptor-Gene and Sexual Function in Middle Aged Women
Acronym: CAG-Libido
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital Muenster (Other); University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 087/13
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Libido; Receptors, Androgen; Polymorphism, Genetic; Androgen Effect
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: All study participants

SUMMARY:
It is known that with increasing age sexual desire is declining in women. Decreasing levels of androgens are believed to have an influence, but cannot explain the loss of libido completely. A possible explanation might be that the effect of the androgen is depending on the functionality of the androgen receptor. It is known that this functionality is genetically determined by the polymorphism of the androgen receptor gene. In the gene there is a varying number of CAG-repeats: the longer the CAG-Repeat, the lower the functionality of the androgen receptor, the lower the effect of the androgens. In this pilot study, the investigators would like to invite 45 healthy heterosexual middle-aged women to the University Hospital of Bern, where they answer questionnaires about their sexual function and where they give a blood sample to assess the testosterone serum levels and the genetically determined androgen receptor subtype.

The investigators believe that lower androgen levels and/or longer CAG-repeats in the androgen receptor gene are related to lower libido scores in healthy middle-aged women.

DETAILED DESCRIPTION:
Background

It is known that with increasing age sexual desire is declining in women. Multiple factors are being discussed to have an influence on this topic, such as cultural, individual and biological factors. Decreasing levels of sexual hormones and specifically androgens are believed to have an influence, hence a lot of women benefit from a testosterone replacement therapy. Yet the sole decline of androgen levels with inclining age cannot explain the loss of libido completely.

A possible further factor might be the androgen receptor: It is known that the effect of the androgen in its target cells is depending on the functionality of the androgen receptor. This functionality is genetically determined by the polymorphism of the androgen receptor gene: In the gene there is a sequence with a varying number of CAG-repeats. This CAG-repeat is coding for a polyglutamine stretch in the androgen receptor which is responsible for the binding of co-activator proteins. The better these co-activator proteins are bound to the androgen receptor, the better the transcriptional activity of the latter. Previous studies have shown that the longer the CAG-Repeat, the weaker the binding of co-activator proteins, the lower the functionality of the receptor and therefore the lower the effects of the androgen on the target cell. Given this circumstances the same level of androgen can have different effects in two individuals.

Objective

In this pilot study, the investigators would like to correlate the testosterone serum levels, the functionality of the androgen receptor and the libido in 45 healthy, heterosexual middle-aged women.

Methods

45 healthy middle-aged women are being recruited and are being invited to come to the University Hospital in Berne. Here they will answer standardised questionnaires about their sexual function and libido and will give a blood sample to measure all the relevant parameters (fasting, premenopausal women: 1.-5. day of cycle): Total Testosterone, SHBG, Estrogen, DHEAS, FSH, LH, CAG repeats of the androgen receptor gene, TSH, fT3, fT4, Prolactin, Ferritin, CRP, Hemoglobin.

A statistician will then assess the collected data. No interventions are planned.

The following collaborators are providing support for this study: Dr. rer. nat. Ulrich Stefenelli, Würzburg, Germany, and Dr. med. Stefan Schmid, Rheinfelden, Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Healthy
* Heterosexual
* Aged 45-65
* Written Informed Consent
* Living since at least 1 year in a relationship
* Ready to answer questionnaires about their sexual function
* Ready to give a blood sample
* German speaking

Exclusion Criteria

* Serious diseases such as Cancer, Parkinsons Disease, Multiple Sclerosis, Diabetes mellitus
* Sexual Abuse in personal history
* Thyroid dysfunction
* Substance abuse (>1pack/cigarettes per day, alcohol, drugs)
* Psychiatric diseases in personal history
* Acute stressful life event
* Libido affecting diseases such as dyspareunia, vaginism, orgasm disorders, urine incontinence
* Medication with the following substances in the past 8 weeks before day of visit:
* Systemic corticoids
* Blood pressure medication with beta-blockers, spironolactone, thiazide diuretics
* Psychotropic medication such as antidepressants, benzodiazepins, antiepileptics, antipsychotics (1st generation)
* Opioid analgetics
* Hormonal contraceptives
* Libido stimulating medication such as androgens (Testosterone, Dehydroepiandrostendionsulfate, Dihydrotestosterone and PDE5-Inhibitants
* Antiandrogens

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A community sample of 45 healthy heterosexual women, aged 45-65.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
2 Subscores of the Female Sexual Function Index (FSFI): Satisfaction and Desire | 1 Day of visit

SECONDARY OUTCOMES:
Other 4 Subscores of the FSFI: Arousal, Lubrication, Orgasm and Pain | 1 Day of visit
CAG-repeats of the androgen receptor gene | 1 Day of visit
Testosterone serum levels | 1 Day of visit
Androgenity score | 1 Day of visit
  Calculated from Gender-specific Index of Testosterone serum levels, CAG repeats and libido scores
Other influences on libido in middle aged women | 1 Day of visit

CONTACTS AND LOCATIONS:
Overall Officials: Petra Stute, PD Dr. med., Principal Investigator — Clinic for Gynaecology and Obstetrics, Insel University Hospital Bern, Switzerland
Locations (1):
- Dep. of gynaecological Endocrinology and reproduction medicine, Clinic for Gynaecology and Obstetrics, Bern University Hospital, Bern, Switzerland